CLINICAL TRIAL: NCT04223323
Title: SNACKing Study: Effects of Snacking on the Gastrointestinal Microbiota and Metabolism
Brief Title: Effects of Almond Consumption on the Human Gastrointestinal Microbiota and Metabolic Health
Acronym: SNACKing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20154
Record Dates: First submitted 2019-11-12; First posted 2020-01-10 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Overweight and Obesity
Keywords: Almond; Gastrointestinal microbiota; Metabolic health; Bile acid profiles
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention arm consists of daily consumption of the investigator's intervention snack over the course of 12 weeks.
  Interventions: Dietary Supplement: Almonds
- Isocaloric Control (Placebo Comparator): The control arm consists of daily consumption of an isocaloric snack over the course of 12 weeks.
  Interventions: Dietary Supplement: Pretzels

INTERVENTIONS:
Dietary Supplement: Almonds — Participants in the intervention group will consume 2oz of almonds daily over the course of 12 weeks.
  Arms: Intervention
Dietary Supplement: Pretzels — Participants in the control group will consume an isocaloric amount of pretzels daily over the course of 12 weeks.
  Arms: Isocaloric Control

SUMMARY:
The proposed work will investigate the effect of almond consumption as a snack on human gastrointestinal microbiota and on metabolic health.

DETAILED DESCRIPTION:
This study is a randomized, controlled, investigator-blinded, parallel arm design with two treatment conditions. There will be a phone screening, in person pre-intervention testing, a one-week baseline period devoid of all nuts and seeds followed by a 12-week intervention period, and a post-testing appointment. Participants will be randomized to consume almonds or isocaloric snack for 12 weeks. Participants will provide stool samples during baseline testing and during the 12th week of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Males & Females
* 30-60 years of age
* BMI 25-34.9 kg/m^2
* Ability to drop off fecal sample within 15 minutes of defecation

Exclusion Criteria:

* Physician diagnosed metabolic or gastrointestinal diseases
* Fasting blood glucose >126 mg/dL
* Blood pressure >160/100 mm Hg
* Anemia
* Elevation in serum transaminases (i.e. >3 times the upper limit of normal)
* Evidence of liver disease, including primary biliary cirrhosis or gallbladder disease, constipation
* Currently taking lipid-lowering medications, oral hypoglycemic agents, or insulin, or medications known to impact bowel function.
* Pregnant, breastfeeding or postmenopausal
* Smoker, tobacco use
* Allergic to nuts
* Consume > 2 alcoholic beverages/day
* Abuse drugs
* Have had > 5% weight change in the past month or > 10% change in the past year
* Have taken antibiotics during the previous 2 months
* Unable to consume the experimental treatments (almonds or pretzels)
* Bariatric surgery
* Gallbladder removal
* Allergic to lidocaine or other topical anesthetics

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Changes in gastrointestinal microbiota composition | Baseline & 12-week mark
  Determine the impact of daily consumption of almonds on the gastrointestinal microbiota compared to control (pretzels) by sequencing the V4 region of the 16S rRNA gene in fecal samples.
Changes in abundance of fecal Roseburia spp | Baseline & 12-week mark
  Determine the impact of daily consumption of almonds on the abundance of Roseburia spp. compared to control (pretzels) by using quantitative real-time PCR.
Changes in abundance of fecal Butyryl CoA: Acetate CoA transferase | Baseline & 12-week mark
  Determine the impact of daily consumption of almonds on the abundance of Butyryl CoA: Acetate CoA transferase gene compared to control (pretzels) by using quantitative real-time PCR.
Changes in gastrointestinal microbial-derived metabolite concentrations | Baseline & 12-week mark
  Determine the impact of daily consumption of almonds on the concentration of microbial-derived metabolites compared to control (pretzels) by using gas-liquid chromatography. These metabolites include butyrate and secondary bile acids.

SECONDARY OUTCOMES:
Changes in liver fat | Baseline & 12-week mark
  Determine the impact of daily consumption of almonds on liver fat percentages compared to control (pretzels) by quantitative liver ultrasound.
Changes in glycemic control. | Baseline & 12-week mark
  Determine the impact on oral glucose tolerance within intervention (almond) and control (pretzel) groups by using a mixed meal tolerance test.
Changes in secondary measures of gastrointestinal health. | Baseline & 12-week mark
  Determine the impact of daily consumption of almonds on gastrointestinal health compared to control (pretzels) by measuring fecal pH; other microbial fermentation end products and microbial-derived bile acids using gas-liquid chromatography; and alpha- and beta- diversity measures of the gut microbiota community structure using 16S microbiota analyses.

OTHER OUTCOMES:
Changes in markers of systemic inflammation & metabolism | Baseline & 12-week mark
  Determine the impact of daily consumption of almonds on inflammation and metabolism compared to control (pretzels) by measuring biomarker concentrations with ELISA. Specifically, we will look at TNF, CRP, & LPS-BP (inflammatory) and NEFAs (metabolism).
Changes in adiposity. | Baseline & 12-week mark
  Determine the impact of daily consumption of almonds on adiposity compared to control (pretzels) using a DXA scan.
Changes in subjective measures of gastrointestinal health. | Baseline & 12-week mark
  Determine the impact of daily consumption of almonds on subjective measures of gut health compared to control (pretzels) using stool records. The questionnaire addresses questions related to gastrointestinal health including bloating, flatulence, and stool consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Hannah D Holscher, PhD RD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No